CLINICAL TRIAL: NCT00255398
Title: Kidney Disease Biomarkers
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060020; 06-DK-0020
Record Dates: First submitted 2006-07-07; First posted 2005-11-18 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-12-03

CONDITIONS: Kidney Disease; Glomerular Disease; Idiopathic Nephrotic Syndrome; Focal Segmental Glomerulosclerosis; Collapsing Glomerulopathy
Keywords: Focal Segmental Glomerulosclerosis; Minimal Change Disease; Diabetic Nephropathy; Mass Spectrometry; Proteinuria; Idiopathic Nephrotic Syndrome; Glomerular Disease; FSG; Kidney Disease
MeSH Terms: conditions — Kidney Diseases; Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental; Diabetic Nephropathies; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Kidney Disease Biomarkers

Summary: This study will identify biomarkers (proteins and other molecules in the blood or urine) that may help scientists predict what kidney disease a patient has and whether a given patient would respond to particular therapies. The study will look for biomarkers in the blood and urine of patients with various kidney diseases and study of the effects of angiotensin converting enzyme inhibitors (ACE inhibitors) and angiotensin receptor blockers (ARB) on biomarkers. Blood and urine from healthy volunteers will be studied for comparison.

Healthy people and the following patients may be eligible for this study: adults with diabetic nephropathy 18 years of age and older; children with newly diagnosed clinical idiopathic nephrotic syndrome between 2 and 18 year of age; children and adults with glomerular disease (minimal change disease, focal segmental glomerulosclerosis, or collapsing glomerulopathy).

Participants undergo tests and procedures as follows:

Glomerular Disease: Adults with glomerular disease provide about four to six blood and urine samples over the course of 6 to 12 months. The samples are collected at the time of regularly scheduled visits for the NIH treatment protocol in which they are participating. Children provide only blood samples.

Chronic Kidney Disease: Patients with chronic kidney disease provide a blood and urine sample every 6 months for 3 years or more.

Angiotensin Antagonism: Patients with chronic kidney disease who are taking ACE inhibitors or ARBs stop their medicines for 4 weeks, while those who are not taking ACE inhibitors or ARBs begin one of the medicines. In general, patients just starting on the medications continue them after the study is completed, since they are beneficial for chronic kidney disease.

* Medication withdrawal group: Patients come to NIH for 2 successive days at the beginning of the study for blood and urine tests (including one 24-hour urine collection) and to receive iothalamate (a chemical used to measure kidney function). Iothalamate is delivered over 24 hours through a needle placed in the abdomen (or elsewhere) via a pump similar to pumps that some diabetics use to deliver insulin. Patients then stop taking their ACE inhibitor or ARB medication. They monitor their blood pressure every day and return to NIH after 1, 2 and 4 weeks for blood tests. During week 4, the iothalamate infusion is repeated, and blood and urine samples are collected as at the beginning of the study. Patients then resume taking their ACE inhibitor or ARB once a day with the dose being increased at 2-week intervals. They come to NIH weekly after 1 week and then every other week for blood tests. Four weeks after reaching the highest FDA-recommended dose of medication tolerated, the iothalamate infusion and blood and urine collections are repeated.
* Medication induction group: At the beginning of the study, patients have the iothalamate infusion and blood and urine collections described above and then begin to take either an ACE inhibitor or ARB. The dose is increased after 2 weeks. Patients monitor their blood pressure every day. After being on the highest dose for 4 weeks, patients repeat the iothalamate infusion and blood and urine collections. The study is then complete and they are provided a 2-month supply of medicine to take home.

Information is gathered on symptoms, treatments, and results of past laboratory tests of all patients. Healthy volunteers provide blood and urine sample collections every month or every other month for up to four collections to be used for biomarker studies and the screen for common chronic diseases.

DETAILED DESCRIPTION:
There is a pressing need to develop biomarkers for renal disease, which might assist in diagnosis and prognosis and might provide endpoints for clinical trials of drugs designed to slow progression of renal insufficiency. We propose to study potential biomarkers in five populations. First, we will study remittive therapy for glomerular disease (sample size up to 40), enrolling children with idiopathic nephrotic syndrome (N=20) and adults with minimal change, focal segmental glomerulosclerosis, and collapsing glomerulopathy (N=20). We will collect periodic urine samples as these patients receive remittive therapy with glucocorticoids or other agents. We will also study up to 10 healthy adult volunteers. We will carry out targeted urine proteomic studies, measuring levels of glomerular cell markers and cytokines, and we will profile urine proteins using mass spectrometry. Our goals are to identify markers of particular disease entities and of steroid responsiveness and to explore whether biomarkers contribute to the histologic sub-classification of these diseases. Second, we will study up to 40 adults with progressive chronic kidney disease of various etiologies and glomerular filtration rate <60 ml/min/1.73m2. We will study blood and urine samples, using both targeted and profiling approaches. Our goal is to identify biomarkers that correlate with progressive loss of glomerular filtration function, which is a functional correlate of progressive renal fibrosis. Third, we will study up to 40 adults, primarily with diabetic nephropathy, who start or stop angiotensin antagonist therapy (angiotensin converting enzyme inhibitors or angiotensin receptor blockers) and compare urine proteomic profiles on therapy and off therapy (4 week interval). Our goal is to identify potential biomarkers that correlate with the beneficial anti-fibrotic effects of these agents. Fourth, we wish to define possible sex differences in urine exosome proteins, obtained from healthy volunteers, who are hospitalized for six days for administration of a standard diet and collection of research urine samples. Fifth, we wish to determine whether salt intake influences urine exosome proteins, obtained from healthy volunteers. These subjects will be hospitalized for 12 days during which time they will be placed sequentially on a high salt diet and a low salt diet, with collection of research urine samples and blood pressure monitoring. Proteomic analysis in these studies will take several approaches, including mass spectrometry of urinary peptides, analysis of urinary exosomes, and immunologic detection and quantification of candidate proteins in urine and blood.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Children with newly diagnosed clinical idiopathic nephrotic syndrome between the ages of 2-18 years.
  2. Children with previously diagnosed clinical idiopathic nephrotic syndrome between the age of 2-18 years at the time of diagnosis who sustain a relapse of nephrotic syndrome while off steroid therapy. A relapse is defined as a urine protein level of 2+ (100mg/dl) or greater on a first morning urine sample for 3 consecutive days. While a quantitative urine protein/creatinine ratio is more precise, this semi-quantitative definition accords with pediatric practice. Relapses will be treated according to standard clinical practice.
  3. Children and adults who participate in NIH trials of remittive therapy for MCD/FSGS/CG (e.g. Podocyte dexamethasone or Retinoids for podocyte disease) will be eligible.
  4. Also, we will study up to 10 healthy adult volunteers.

EXCLUSION CRITERIA:

1. IN CHILDREN, ANY OF THE FOLLOWING

   1. Age less than 2 years. The rationale for excluding children under the age of 2 yr is that nephrotic syndrome is unusual in this age group and may have etiologies other than MCD and FSGS
   2. Uncontrolled hypertension (a systolic or diastolic which is greater than 95% population mean for child s age and sex, while receiving therapy), azotemia (serum creatinine greater than 1.5mg/dL), gross hematuria at the time of presentation (clinical markers of primary or secondary GN).
   3. Hypocomplementemia, positive ANA, anti-DS DNA, ASO, anti-DNase B, MPO, PR-3, Hepatitis B and C and HIV serologies.
2. In children or adults:

   1. Clinical contra-indications to steroid therapy.
   2. The presence of medical conditions that might interfere with the interpretation of results, such as cancer, diabetes, or a long history of hypertension.
3. Healthy adult volunteers:

   1. age greater than 18 yrs; no history of hypertension, diabetes, or other chronic illness that might complicate interpretation of the results; not taking prescription medication.

      CKD PROGRESSION STUDY:

      INCLUSION CRITERIA:
      1. Renal biopsy diagnosis of glomerular disease or interstitial nephritis or clinical diagnosis of diabetic nephropathy.
      2. Mild or moderate renal insufficiency, defined as eGFR less than 60 ml/min/1.73m(2) but greater than 30 ml/min/1.73m(2).

      EXCLUSION CRITERIA:

      1) The presence of medical conditions that might interfere with the interpretation of results, such as cancer.

      ANGIOTENSIN ANTAGONISM STUDY:

      INCLUSION CRITERIA:
      1. Adults greater than 18 years old. Few children have diabetic nephropathy and the frequent blood draws would be problematic for children.
      2. Type 1 or Type 2 diabetes. Later studies will be expanded to other glomerular diseases.
      3. Urinary albumin/creatinine ratio greater than 30 mg/g. The rationale is to include patients with macroproteinuria and patients with microalbuminuria.
      4. Estimated GFR greater than 30 mL/min/1.73m(2). The rationale is to exclude patients with severe CKD.

      EXCLUSION CRITERIA:
      1. Allergy to ACE inhibitor or ARB
      2. Current or planned pregnancy; urine HCG performed at start of study and on the day of iothalamate infusion.
      3. Serum potassium greater than 5.0 mEq/L off angiotensin antagonist therapy
      4. The presence of medical conditions which would make interpretation of results difficult such as cancer.
      5. History of iodine allergy or severe asthma (history of emergency department visit or hospitalization).

      SEX DIFFERENCES IN URINARY EXOSOME PROTEINS:

      INCLUSION CRITERIA:
      1. Age 18-30; Young adults are less likely to have undetected chronic renal disease.
      2. BMI 18-27.5 kg/m(2); Obesity may alter renal function.
      3. BP consistently less than 130/80; Pre-hypertension or hypertension may affect the kidney.

      EXCLUSION CRITERIA:
      1. Any chronic illness that might interfere with interpretation of the study; certain illnesses that do not require therapy may be consistent with inclusion, including mild asthma or psychiatric illness.
      2. Cancer other than non-melanoma skin cancer in the past 5 years.
      3. Need for any chronic or intermittent medication other than acetaminophen.
      4. Women: amenorrhea, irregular menses, menstrual cycles less than 26 days or greater than 32 days, or use of contraceptive hormones (unwilling or unable to switch to non-hormonal means of contraception); Irregular cycle may be non-ovulatory and associated with abnormal sex hormone profiles, which will complicate data interpretation.
      5. Use of nicotine or illicit drugs.
      6. Febrile illness or urinary tract infection: postpone admission one week or more.

      SALT INTAKE AND BLOOD PRESSURE RESPONSES IN URINARY EXOSOMES:

      INCLUSION CRITERIA:
      1. Men Age 18-35
      2. BMI 18-25 kg/m(2)
      3. BP consistently less than 130/80

      EXCLUSION CRITERIA:
      1. Any chronic illness that might interfere with interpretation of the study; certain illnesses that do not require therapy may be consistent with inclusion, including mild asthma or psychiatric illness
      2. Cancer other than non-melanoma skin cancer in the past 5 years
      3. Need for any chronic or intermittent medication other than acetaminophen
      4. Use of nicotine or illicit drug
      5. Febrile illness or urinary tract infection: postpone admission one week or more

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-11-10; Study Completion 2014-12-03

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Kopp, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barisoni L, Kopp JB. Modulation of podocyte phenotype in collapsing glomerulopathies. Microsc Res Tech. 2002 May 15;57(4):254-62. doi: 10.1002/jemt.10084. PMID 12012394
- [Background] Savin VJ, McCarthy ET, Sharma M. Permeability factors in focal segmental glomerulosclerosis. Semin Nephrol. 2003 Mar;23(2):147-60. doi: 10.1053/snep.2003.50024. PMID 12704575
- [Background] Hortin GL, Meilinger B, Drake SK. Size-selective extraction of peptides from urine for mass spectrometric analysis. Clin Chem. 2004 Jun;50(6):1092-5. doi: 10.1373/clinchem.2003.030742. No abstract available. PMID 15161733